CLINICAL TRIAL: NCT00883025
Title: Correlation Between Friedman Classification Ande ApneaHypopnea Index in a Population With OSAS
Brief Title: Correlation Between Friedman Classification and the Apnea Hypopnea Index (AIH) in a Population With Obstructive Sleep Apnea Syndrome (OSAS)
Acronym: FriedmAIH
Status: Completed | Type: Observational
Sponsor: Irmandade da Santa Casa de Misericoridia de Limeira (Other)
Collaborators: Hospital Dia (Unknown)
Responsible Party: Marcos Marques Rodrigues, Irmandade da Santa Casa de Misericoridia de Limeira
Other Study IDs: CEP ISCML 113/08; FriedmanAIH
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Friedman Classification; Apnea-Hypopnea Index; Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: OSAS patients
- 2: no OSAS Patient

SUMMARY:
Introduction:

OSAS is an important disease in the actual medic scene. It is important for correlation with chronic cardiovascular disease that leaves an increase in morbimortality and socioeconomic disability to patients with apnea.

Objectives:

Determinate the correlation between Friedman Classification and the obstructive sleep apnea syndrome (OSAS) gravity through AHI (Apnea Hypopnea Index) in patients with OSAS for surgical indication and evaluation.

Materials and Methods:

The investigators evaluated and classified 84 patients, in the scale of Epworth, Friedman and how much the gravity of the SAHOS for the AHI.

ELIGIBILITY:
Inclusion Criteria:

* Not exhibiting any exclusion criteria
* Age > 21 years

Exclusion Criteria:

* Nasal tumor
* BMI > 40
* No acceptance of study
* Nasal poliposis

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of Ambulatory of Sleep Respiratory Disorders of Santa Casa de Limeira
Enrollment: 147 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Friedman Classification | one year

SECONDARY OUTCOMES:
Apnea-Hypopnea Index | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Dia, Limeira, São Paulo, Brazil

REFERENCES:
- [Derived] Rodrigues MM, Dibbern RS, Santos VJ, Passeri LA. Influence of obesity on the correlation between laryngopharyngeal reflux and obstructive sleep apnea. Braz J Otorhinolaryngol. 2014 Jan-Feb;80(1):5-10. doi: 10.5935/1808-8694.20140004. English, Portuguese. PMID 24626885